CLINICAL TRIAL: NCT04773067
Title: A Phase II, Placebo-controlled, Randomized, Observer-blind Study to Evaluate the Immunogenicity, Safety, and Tolerability of UB-612 Vaccine Against COVID-19 in Adolescent, Younger and Elderly Adult Volunteers
Brief Title: A Study to Evaluate UB-612 COVID-19 Vaccine in Adolescent, Younger and Elderly Adult Volunteers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Under the limited resources, to re-plan the ongoing clinical trials of this product.
Sponsor: United Biomedical Inc., Asia (Industry)
Collaborators: Vaxxinity, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V-205
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — UB-612 COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UB-612 (Experimental): A proprietary high-precision designer S1-RBD protein based vaccine incorporating Th/CTL peptides to activate T cells.
  Interventions: Biological: UB-612
- Placebo (Placebo Comparator): Normal saline 0.9%.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: UB-612 — Around 3300 adult subjects and 330 adolescent subjects will receive 2 doses of 100 µg UB-612 vaccine. The subjects will be invited to have the 3rd dose after unblinded.
  Arms: UB-612
Biological: Placebo — Around 550 adult subjects and 55 adolescent subjects will receive 2 doses of normal saline 0.9%.
  Arms: Placebo

SUMMARY:
This is a phase II, observer-blind, multiple-centre, randomized, placebo-controlled study to evaluate the immunogenicity, safety, tolerability and lot consistency of 2 doses of UB-612 vaccine in adolescent, younger and elderly adults. Around 3850 adult subjects will be randomized to be composed of the core group, while around 385 adolescents will be randomized to be the supplementary group. Subjects will be unblinded at Visit 5, and subjects in the vaccine group will be encouraged to have 3rd dose of vaccination.

DETAILED DESCRIPTION:
This clinical study will be consisted of 7 clinical visits and one long-term follow-up visit. Subjects will also be unblinded at Visit 5, subjects in placebo group will withdraw from the study and subjects in vaccine group will be encouraged to have 3rd dose of vaccination (Day 197~Day 242) at Visit 6. Those who received 3rd dose will have Visit 7 (14 days after Visit 6) to check the booster effect. After Day 197, subjects will enter the long-term follow-up with a safety call bi-monthly.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female between the age of 12 to 85 years at time of enrolment.
* Women of childbearing potential and men must agree to practice medically effective contraception from first vaccination until 3 months after the last vaccination.
* Able to understand the content and possible risks of informed consent and willing to sign the Informed Consent Form (ICF).
* Able to understand and agrees to comply with all study procedures and be available for all study visits.
* Ear temperature ≤ 38.0°C.
* Healthy participants who are determined by medical history, physical examination, and clinical judgment of the investigator to be eligible for inclusion in the study. In the investigator's clinical judgement, participant may have a stable and well-controlled comorbidity associated with an increased risk of progression to severe COVID-19.

Exclusion Criteria:

* History of anaphylaxis, urticarial, or other significant adverse reaction requiring medical intervention after receipt of a vaccine.
* Female who is pregnant or positive in pregnancy test at screening or just prior to each vaccination administration.
* Female who is breast-feeding or plans to breastfeed from the time of the first vaccination through 60 days after the last vaccination.
* Any acute illness, as determined by the study investigator 3 days before first vaccination (these subjects can be re-scheduled).
* Any major surgery one month before first vaccination (these subjects can be -rescheduled).
* Known HIV antibody positive.
* Known active hepatitis B and hepatitis C disease.
* Previous exposure to SARS-CoV-2 or receipt of an investigational or licensed product for the prevention of COVID-19, MERS or SARS.
* Have history of Guillain-Barre syndrome.
* Subjects who take part in another clinical study within 12 weeks prior to the day of informed consent.
* Immune deficiency/disorder, whether due to genetic defect, immunodeficiency disease or immunosuppressive therapy.
* Subjects who plan to or are undergoing anti-cancer therapy.
* Platelet disorder or other bleeding disorder may cause injection contraindication.
* Prior chronic administration of immunosuppressant or corticosteroids, cytotoxic treatment in last 6 months before first vaccination.
* Prior administration of immunoglobulins and/or any blood products in last 4 months before first vaccination.
* Receipt of any seasonal or pandemic influenza vaccine within 14 days, or any other non-study vaccine within 28 days, before study intervention administration.
* Anticipated receipt of any seasonal or pandemic influenza vaccine within 14 days, or any other nonstudy vaccine within 28 days, after study intervention administration.
* Receipt of short-term (<14 days) systemic corticosteroids. Study intervention administration should be delayed until systemic corticosteroid use has been discontinued for at least 28 days. Inhaled/nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
* Loss or donation of blood over 500 mL within 3 months prior to Screening Visit or intention to donate blood or blood products for transfusion during the study.
* Any medical disease or condition that, in the opinion of the study investigator, may confound the results of the study or pose an additional risk to the subjects by their participation in the study.
* Employees at the investigator's site, of the Sponsor or the contract research organization (CRO) who directly involved in the conduct of the study.

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3877 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) of SARS-CoV-2 neutralizaing antibody | Day 57
  Immunogenicity evaluation
Seroconversion rate (SCR) of SARS-CoV-2 neutralizing antibody | Day 57
  Immunogenicity evaluation
Local reactions and systemic events | Up to 7 days following each dose
  Safety evaluation
Unsolicited adverse events | Day 1 to Day 57
  Safety evaluation
Medically attend adverse events (MAAEs), serious adverse events (SAEs), adverse event of special interests (AESIs) and antibody dependent enhancements (ADEs) | Day 1 to Day 365
  Safety evaluation

SECONDARY OUTCOMES:
SCR of anti-S1-RBD antibody | Day 57
  Immunogenicity evaluation
GMT of SARS-CoV-2 neutralizing antibody | Day 197 and 365
  Immunogenicity evaluation
GMT of anti-S1-RBD antibody | Day 57, 197 and 365
  Immunogenicity evaluation
Geometric mean fold increase in SARS-CoV-2 neutralizing antibody and antigen-specific antibody (Anti-S1-RBD) | Day 57, 197 and 365
  Immunogenicity evaluation
Lot consistency by comparisons of GMT of SARS-CoV-2 neutralizing antibody | Day 57
  Evaluation of lot to lot consistency

OTHER OUTCOMES:
Antigen-specific interferon-gamma (IFN-γ) and IL-4 production measured by ELISpot | Day 57 and 14 days post 3rd dose
  Evaluation of T cell function induced by UB-612
CD4+ and CD8+ T cell responses measured by flow cytometric assays | Day 57 and 14 days post 3rd dose
  Evaluation of T cell function induced by UB-612
GMT of SARS-CoV-2 neutralizing antibody | 14 days post 3rd dose
  Immunogenicity evaluation
GMT of anti-S1-RBD antibody | 14 days post 3rd dose
  Immunogenicity evaluation
Geometric mean fold increase in SARS-CoV-2 neutralizing antibody and anti-S1-RBD antibody | 14 days post 3rd dose
  Immunogenicity evaluation
GMT of SARS-CoV-2 neutralizing antibody and anti-S1-RBD antibody in adolescents | Day 57, Day 197 and Day 365
  Immunogenicity evaluation
SCR of SARS-CoV-2 neutralizing antibody and anti-S1-RBD antibody in adolescents | Day 57
  Immunogenicity evaluation
Geometric mean fold increase in SARS-CoV-2 neutralizing antibody and anti-S1-RBD antibody in adolescents | Day 57, Day 197, and Day 365
  Immunogenicity evaluation
Safety evaluation in adolescents | Day 1 to Day 365
  1. Local reactions and systemic events for up to 7 days following each dose
  2. Unsolicited AEs from Day 1 to Day 57
  3. MAAEs, SAEs, AESIs and ADEs from Day 1 to Day 365
Incidence of COVID-19 cases | Day 1 to Day 365
  COVID-19 incidence per 1000 person-years of follow-up
Antibody against SARS-CoV-2 antigens measured by ELISA | Day 1 to Day 365
  Antigens derived from S2, N and M protein.

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Yi Wang, Ph.D., Study Chair — United Biomedical Inc., Asia
Locations (12):
- Taiwan (12):
  - Changhua Christian Hospital, Changhua
  - Chang-Geng Medical Foundation Kaoshiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang-Geng Medical Foundation Linkou Chang-Geng Memorial Hospital, Taoyuan District

REFERENCES:
- [Derived] Wang CY, Peng WJ, Kuo BS, Ho YH, Wang MS, Yang YT, Chang PY, Shen YH, Hwang KP. Toward a pan-SARS-CoV-2 vaccine targeting conserved epitopes on spike and non-spike proteins for potent, broad and durable immune responses. PLoS Pathog. 2023 Apr 20;19(4):e1010870. doi: 10.1371/journal.ppat.1010870. eCollection 2023 Apr. PMID 37079651
- [Derived] Wang CY, Hwang KP, Kuo HK, Peng WJ, Shen YH, Kuo BS, Huang JH, Liu H, Ho YH, Lin F, Ding S, Liu Z, Wu HT, Huang CT, Lee YJ, Liu MC, Yang YC, Lu PL, Tsai HC, Lee CH, Shi ZY, Liu CE, Liao CH, Chang FY, Chen HC, Wang FD, Hou KL, Cheng J, Wang MS, Yang YT, Chiu HC, Jiang MH, Shih HY, Shen HY, Chang PY, Lan YR, Chen CT, Lin YL, Liang JJ, Liao CC, Chou YC, Morris MK, Hanson CV, Guirakhoo F, Hellerstein M, Yu HJ, King CC, Kemp T, Heppner DG, Monath TP. A multitope SARS-CoV-2 vaccine provides long-lasting B cell and T cell immunity against Delta and Omicron variants. J Clin Invest. 2022 May 16;132(10):e157707. doi: 10.1172/JCI157707. PMID 35316221